CLINICAL TRIAL: NCT05369507
Title: Eliminating HCV in Rural South Carolina With Smart Phone Virtual Care Coordination Deployed in NP Led Mobile Clinics
Brief Title: Eliminating HCV in Rural South Carolina Utilizing NP Led Mobile Clinics and Virtual Care Coordination
Acronym: STAT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00106348
Record Dates: First submitted 2022-05-05; First posted 2022-05-11 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis C; Substance Use Disorders
Keywords: Mobile health; Nurse practitioner; Care coordination; Virtual care coordination; People who inject drugs; Rural health
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: At time of randomization, participant is informed of study group assignment and provided instructions on use of app. Care provider is aware of group assignment as the provider is also using the platform to communicate with participants during course of treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): TAU group will receive standard care coordination efforts by health care team throughout course of HCV treatment
- Virtual Care Coordination (Experimental): Participants will download a mobile phone app (emocha) to facilitate care coordination throughout course of HCV treatment
  Interventions: Behavioral: Virtual Care Coordination

INTERVENTIONS:
Behavioral: Virtual Care Coordination — Participants randomly assigned to the virtual care coordination group will use a mobile app to assist in HCV treatment care coordination.
  Arms: Virtual Care Coordination

SUMMARY:
Up to 150 individuals with current hepatitis C (HCV) will be recruited from mobile health clinics in rural South Carolina - sites will be selected based on HCV prevalence rates and lack of current HCV screening/treatment resources. NPs will provide HCV care through mobile health units. Participants will be randomized (1:1) to either mobile health clinic treatment as usual or virtual care coordination. Virtual care coordination designed to move people along HCV care cascade will be conducted by the Emocha smartphone platform - an adaptable platform designed by emocha to link patients to care. Using quantitative methods, associations between psychosocial factors such as homelessness, mental illness, provider mistrust, poor social support, high levels of shame and stigma with HCV outcomes including SVR will be examined. Investigators hypothesize that SVR rate among the HCV-infected individuals treated (and with follow-up SVR determination) will be 90% with the Clopper-Pearson 95% CI having a width of 13%.

ELIGIBILITY:
Inclusion Criteria:

* Not previously treated with HCV direct-acting antiviral medications OR treatment-experienced and eligible for treatment with sofosbuvir/velpatasvir
* Age 18+
* Willing to be randomized to either emocha versus TAU arms
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
HCV Treatment Initiation Rates | 27 months
  To determine whether treatment initiation rates are higher among patients randomized to Emocha virtual care coordination versus treatment as usual (TAU), among HCV-infected patients enrolled in a NP-led mobile clinic

SECONDARY OUTCOMES:
HCV Treatment Adherence | 12 weeks
  Measured by pharmacy refills
HCV Treatment Completion | 12 weeks
  Measured by 100% completion of 12-week treatment course
Rate of Sustained Virologic Response | 6 months
  Measured by end of treatment SVR labs

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No